CLINICAL TRIAL: NCT00344760
Title: Viral Decay Kinetics During Induction Therapy With or Without the Use of Enfuvirtide in HAART-naÃ-ve Patients With Advanced HIV
Brief Title: A Study to Evaluate of the Efficacy of Enfuvirtide During the Induction Phase of Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-26280
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide; efavirenz; Lamivudine; Tenofovir; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Treatment (Active Comparator): Efavirenz 600mg once daily, Lamivudine 300mg once daily and Tenofovir 300mg once daily
  Interventions: Drug: Efavirenz, lamivudine, and tenofovir
- Standard Treatment Plus Enfuvirtide (Experimental): Efavirenz 600mg once daily, Lamivudine 300mg once daily, Tenofovir 300mg once daily and enfuvirtide 90mg subcutaneously twice a day until the viral load is less than 50copies for 2 consecutive visits or 12 weeks (whichever comes first).
  Interventions: Drug: Enfuvirtide; Drug: Efavirenz, lamivudine, and tenofovir

INTERVENTIONS:
Drug: Enfuvirtide — subcutaneously twice a day
  Other Names: Fuzeon (T-20)
  Arms: Standard Treatment Plus Enfuvirtide
Drug: Efavirenz, lamivudine, and tenofovir — Efavirenz -600mg once daily, lamivudine- 300mg once daily, and tenofovir 300mg once daily
  Other Names: Atripla, Epivir and Viread

SUMMARY:
We hypothesize that using a potent antiretroviral such as Enfuvirtide during the induction phase of HAART therapy will lead to faster clearance of virus and infected cells, and lower number of minority variant HIV-1 strains.

DETAILED DESCRIPTION:
This is an 48 week Phase 4, open label, randomized, prospective, pilot proof of concept study to evaluate the use of Enfuvirtide in an induction/maintenance treatment model. Patients meeting inclusion criteria will be stratified into two groups according to HIV-1 RNA viral loads (less than 300,000 copies/ml and greater than 300,000 copies/ml). Thereafter, patients will be block randomized (the size of each block will be two patients) into one of two treatment arms.

All patients will receive Efavirenz 600mg once a day, Lamivudine 300 mg once a day, and Tenofovir 300mg once a day. After randomization, one half of the patients will receive no additional treatment, while the other half will receive Enfuvirtide 90mg sq BID until the viral load is <50 x 2 consecutive visits or 12 weeks (whichever comes first).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 70 years of age.
2. Sex: Male or Female.
3. Documented HIV-1 seropositive by Western Blot, Elisa, or HIV-1 viral load.
4. Naïve to HAART.
5. Viral load >100,000c/ml.
6. CD4<200c/ml.
7. Volunteers must be willing and able to provide written informed consent to participate in the study.
8. Available for at least 48 weeks of follow-up.

Exclusion Criteria:

1. Volunteers with an acute and clinically significant medical event as determined by the investigator to result in a life expectancy less then 12 months despite ART.
2. Volunteers with current psychiatric illness, alcohol abuse or illicit drug use that in the opinion of the Principal Investigator may interfere with patient's ability to comply with protocol requirements.
3. Renal insufficiency (Estimated Creatinine clearance of <60ml/min.)
4. Patients with malabsorption or severe chronic diarrhea for more than 30 days.
5. Inability to consume adequate oral intake (defined as inability to eat at least 1 meal per day).
6. Current treatment for malignancy other than basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
7. Any other medical condition which, in the opinion of the investigator, might interfere with completion of the study or evaluation of the results.
8. Pregnancy or breastfeeding
9. In a female capable of child bearing, unwillingness to use effective barrier contraception or abstinence
10. Patient who is currently receiving an experimental medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2005-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Time to viral suppression below 50c/ml. | Individual
  The study is 48 weeks long and the time to viraL suppression will vary depending on the subject. Or there is the possibility that they do not supress

SECONDARY OUTCOMES:
Log viral copy/ml decrease over time during phase 1 and phase 2. | Over the 48 week study period
Development of clinical mutations. | Over the 48 week study period
Development of sub-clinical mutations (minority variants) | Over the 48 week study period
Viral suppression (below 50c/ml) at 24 and 48 weeks. | At 24 and 48 weeks
Time to loss of viral response. Loss of viral response defined as: | Over the 48 week study period
Less then 2.0 log decrease in viral load at week 8. | Week 8
Inability to achieve Viral load <50c/ml by week 12. | Week 12
Viral load >50c/ml on 2 consecutive measurements taken 2 weeks apart after viral | Over the 48 week study period
suppression <50c/ml has occurred | Over the 48 week study period
Rate and quantity of HIV-1 proviral DNA decay. | Over the 48 week study period
Safety and tolerability. | Over the 48 week study period

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B Reisler, MD, MPH, Principal Investigator — University of Maryland, School of Medicine, Department of Infectious Disease
Locations (1):
- University of Maryland, Institute of Human Virology, Baltimore, Maryland, United States